CLINICAL TRIAL: NCT00839826
Title: Oral Direct Factor Xa Inhibitor BAY 59-7939 in the Prevention of VTE in Patients Undergoing Total Hip Replacement. ODiXahip - a Phase IIa Dose Escalating Proof of Principle Trial
Brief Title: ODiXahip - a Phase IIa Dose Escalating Proof of Principle Trial
Acronym: ODiXaHip
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10942
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Thromboembolism; Prevention
Keywords: Prevention of Thromboembolism after total hip replacement
MeSH Terms: conditions — Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Active Comparator)
  Interventions: Drug: Enoxaparin
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — 2,5 mg bid,5 mg bid,10mg bid, 20 mg bid, 20 mg tid, 30 mg bid, dose escalation trial
  Arms: Arm 1
Drug: Enoxaparin — 40 mg bid
  Arms: Arm 2

SUMMARY:
Patients undergoing surgery, especially hip and knee surgery, are at high risk for VTE (up to 60 % without prophylaxis). The administration of drugs for thromboprophylaxis, such as heparins, significantly lowers that risk, but heparins have to be applied below the skin (subcutaneously). Additionally, there is a chance of developing a heparin-induced thrombocytopenia (decrease in platelets). Therefore, there is still a need for new agents which are safer and more efficient and which are easier to apply.The purpose of this study is to compare the safety and efficacy of BAY 59-7939 with the safety and efficacy of the licensed drug Enoxaparin. Enoxaparin, a so-called low molecular heparin, is approved and widely used in the area of thromboprophylaxis and will be given once daily subcutaneously.Another important purpose of the study is to find the optimal dose of BAY 59-7939 for thromboprophylaxis after hip replacement surgery. Therefore, there are several dose steps planned.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or above and postmenopausal female patients.
* Patients scheduled for elective primary total hip replacement (cemented or non-cemented prosthesis).
* Patients' written informed consent for participation after receiving detailed written and oral previous information to any study specific procedures.

Exclusion Criteria:

* DVT or PE within the previous 6 months prior to study entry.
* Myocardial infarction (MI) or cerebrovascular attack (CVA), TIA or ischaemic stroke within the last 6 months prior to study entry.
* History of heparin-induced thrombocytopenia, allergy to heparins.
* Intracerebral or intraocular bleeding within the last 6 months prior to study entry.
* History of gastrointestinal disease with gastrointestinal bleeding within the last 6 months prior to the study.
* History or presence of gastrointestinal disease which could result in an impaired absorption of the study drug
* Amputation of one leg.Related to current symptoms or findings
* Heart insufficiency NYHA III-IV.
* Congenital or acquired haemorrhagic diathesis (PT INR/aPTT not within normal limits).
* Thrombocytopenia (platelets < 50.000/µl).
* Macroscopic haematuria.
* Allergy to contrast media.
* Severe hypertension (SBP > 200mmHg, DBP > 100 mmHg).
* Impaired liver function (transaminases > 2 x ULN).
* Impaired renal function (serum creatinine > 1.5 x ULN).
* Active malignant disease.
* Presence of active peptic ulcer or gastrointestinal disease with increased risk of gastrointestinal bleeding.
* Body weight < 45 kg.
* Drug- or alcohol abuse.
* Related to current treatment

  * Therapy with oral anticoagulants (e.g. phenprocoumon, warfarin-sodium).
  * Therapy with acetylic salicylic acid or other thrombocyte aggregation inhibitors (e.g. clopidogrel, dipyridamole and ticlopidine) should be stopped one week before enrolment
  * Treatment with heparins or Factor Xa Inhibitors other than study medication.
  * All other drugs influencing coagulation, (exception: NSAIDs with half life < 17 hrs will be allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2002-12; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is a composite endpoint of: - Any DVT (proximal and/or distal) and - Non fatal PE and - Death from all causes. The primary endpoint will be evaluated 5 - 9 days after surgery. | Assymptomatic DVT will be measured 5-9 days after surgery Symptomatc DVT , non-fatal PE and Death from all causes will be measured 41 days after surgery

SECONDARY OUTCOMES:
Incidence of DVTs (total, proximal, distal) | will be evaluated 5 - 9 days after surgery.
Incidence of symptomatic VTEs | 41 days after surgery
The composite endpoint that results from the primary endpoint by using alternative definition of deaths (i.e. VTE related death) | 41 days after surgery
Incidence of symptomatic VTEs (total, PE, DVT) within 30 days after stop of treatment with the study drug. | 41 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (39):
- Austria (3):
  - Wiener Neustadt, Lower Austria
  - Linz, Upper Austria
  - Vienna, Vienna
- Belgium (4):
  - Baudour
  - Brussels
  - Ghent
  - Huy
- Denmark (4):
  - Hellerup
  - Herlev
  - Hørsholm
  - Silkeborg
- France (3):
  - Amiens
  - Lille
  - Nancy
- Germany (6):
  - Rheinfelden, Baden-Wurttemberg
  - Fürth, Bavaria
  - Garmisch-Partenkirchen, Bavaria
  - Frankfurt am Main, Hesse
  - Dresden, Saxony
  - Berlin, State of Berlin
- Israel (4):
  - Haifa, Israel
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin
- Netherlands (2):
  - Amersfoort
  - Zwolle
- Norway (3):
  - Notodden
  - Oslo
  - Rjukan
- Poland (6):
  - Bialystok
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
- Sweden (3):
  - Gothenburg
  - Jönköping
  - Kungälv
- London, Greater London, United Kingdom